CLINICAL TRIAL: NCT03986242
Title: Vibration Rolling, Non- Vibration Rolling,and Static Stretching for Delayed-onset Muscle Soreness on Physiological Changes and Recovery of Athletic Performance in Runners
Brief Title: Vibration Rolling, Non- Vibration Rolling,and Static Stretching for Delayed-onset Muscle Soreness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: KMUHIRB-F(I)-20180006
Record Dates: First submitted 2019-06-06; First posted 2019-06-14 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-06

CONDITIONS: Delayed-onset Muscle Soreness
Keywords: Delayed-onset muscle soreness; vibration therapy; foam roller; stretching exercise; recovery; performance
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- static stretchin (Experimental): Static extremity muscles of the lower extremities, including: gluteal muscles (major muscle group: gluteus maximus), anterior thigh muscles (strand rectus, medial femoral muscle, lateral femoral muscle, medial femoral muscle), posterior thigh muscles (main muscle) Group: semimembranosus, semitendinosus, biceps femoris), anterior muscles of the calf (anterior tibialis anterior muscle, extensor muscle), and posterior muscles of the calf (gastrocnemius, soleus muscle). 4 groups per muscle group, 30 seconds/group
  Interventions: Other: static stretching
- non- vibration rolling (Experimental): Lower limb part. Such as: gluteal muscle (main muscle group: gluteus maximus), anterior thigh muscle group (straight rectus, medial femoral muscle, lateral femoral muscle, femoral intermediate muscle), posterior thigh muscle group (main muscle group: semimembranosus, Semitendinosus, biceps femoris), anterior muscles of the calf (anterior tibialis anterior muscle, extensor muscle), and posterior muscles of the calf (gastrocnemius, soleus muscle). Each leg of each pair performs 30 seconds/group for a total of 4 groups for a total time of 20 minutes.
  Interventions: Device: rolling
- Vibration rolling (Experimental): Lower limb part. Such as: gluteal muscle (main muscle group: gluteus maximus), anterior thigh muscle group (straight rectus, medial femoral muscle, lateral femoral muscle, femoral intermediate muscle), posterior thigh muscle group (main muscle group: semimembranosus, Semitendinosus, biceps femoris), anterior muscles of the calf (anterior tibialis anterior muscle, extensor muscle), and posterior muscles of the calf (gastrocnemius, soleus muscle). Each muscle group of each foot performs 30 seconds/group, a total of 4 groups, the vibration frequency is 28 Hz, and the total time is 20 minutes.
  Interventions: Device: Vibration rolling

INTERVENTIONS:
Device: rolling — use non- vibration rolling and the total time is 20 minutes.
  Arms: non- vibration rolling
Device: Vibration rolling — use Vibration rolling the vibration frequency is 28 Hz, and the total time is 20 minutes.
  Arms: Vibration rolling
Other: static stretching — static stretching and the total time is 20 minutes.
  Arms: static stretchin

SUMMARY:
Delayed-onset muscle soreness (DOMS) is an acute micro-trauma or inflammatory response experienced in the most runners; and, it concurrently impairs athletic performance and may increase the risk of sports injury. Alleviating the symptoms of DOMS strategies are various; however, the specific recovery way remains unconcluded. Furthermore, few studies have investigated the effects of vibrating roller on alleviating the symptoms of DOMS and understand the biochemical changes in response to recovery of athletic performance. Therefore, this study hypothesizes that vibration rolling (VR) could provide a self-myofascial release. Meanwhile, vibration exercise could transmit vibration to specific muscle groups to decrease inflammation in corresponding to reduce muscular pain. Therefore, it could offer positive effects including improvements of flexibility, muscle stiffness, visual analog scale (VAS) for pain, jump, and dynamic balance.

DETAILED DESCRIPTION:
Background: Delayed-onset muscle soreness (DOMS) is an acute micro-trauma or inflammatory response experienced in the most runners; and, it concurrently impairs athletic performance and may increase risk of sports injury. Alleviating the symptoms of DOMS strategies are various; however, the specific recovery way remains unconcluded. Furthermore, few studies have investigated that the effects of vibrating roller on alleviating the symptoms of DOMS, and understand the biochemical changes in response to recovery of athletic performance. Therefore, this study hypothesizes that vibration rolling (VR) could provide self-myofascia release. Meanwhile, vibration exercise could tramsit vibration to speific muscle groups to decrease inflammation in corresponding to reduce muscular pain. Therefore, it could offer positve effects including improvements of flexability, muscle stiffness, visual analog scale (VAS) for pain, jmup, and dynmaic balance. Purpose: To investigate VR, non-vibration rolling (NVR), and static stretching for DOMS on physiological changes and recovery of athletic performance in runners. Methods: Thirty healthy and recreationally adult runners will be voluntarily recruited in the experiment. Participant will be induced DOMS on the treadmill exercise firstly. Next, participants will be matched up and randomly assigned to the VR group, NVR group or static stretching group treatment. Each participant will be instructed to 20-minutes treatment on bilateral muscles including gluteus, anterior, and posterior thighs as well as anterior, and posterior legs. All subjects will receive blood analysis (leukocyte, lymphocyte, creatine kinase, c-reactive protein, interleukin-6) and perform flexibility muscular stiffness, VAS for pain, counter movement jump, Y balance tests on lower limb before exercise and after 24hour and 48 hour interventions. Expected outcomes: VR could effectively alleviate the symptoms of DOMS including decreasing inflammatory biochemical values, decreasing muscular stiffness, reducing muscular pain, and increasing flexibility and jump ability as well as improving dynamic balance on lower limb. This data may provide in alleviating the symptoms of DOMS to healthy populations, athletes, and medical team members.

Key Words: Delayed-onset muscle soreness, vibration therapy, foam roller, stretching exercise, recovery, performance

ELIGIBILITY:
Inclusion Criteria:

* Recruit runners of regular sports ages 20-40

Exclusion Criteria:

* Less than 3 athletes per week.
* Cardiovascular disease.
* History of asthma.
* Musculoskeletal injury within 6 months.
* Previous fracture surgery.
* Neurological symptoms.
* Taking anti-inflammatory drugs.
* Taking high blood pressure and diabetes.
* Bad habits such as smoking, drinking.
* Not being able to cooperate with time detection.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2018-11-23 (Actual); Primary Completion 2019-06-06 (Actual); Study Completion 2019-06-06 (Actual)

PRIMARY OUTCOMES:
C-reactive protein | Change from baseline at 3 days
  Mainly used as an indicator of inflammation
Interleukin-6 | Change from baseline at 3 days
  Used as an indicator of inflammation

SECONDARY OUTCOMES:
Flexibility | Change from baseline at 3 days
  Sports performance by range of motion (unit=degree). Popliteal angle test to test the range of motion the hamstring. =>Amount of knee extension with hip flexed at 90º
  Ely's test to test the range of motion the rectus femoris.
  =>The therapist is standing next to the patient, at the side of the leg that will be tested.
  One hand should be on the lower back, the other holding the leg at the heel. Passively flex the knee in a rapid fashion. The heel should touch the buttocks. Test both sides for comparison. The test is positive when the heel cannot touch the buttocks, the hip of the tested side rises up from the table, the patient feels pain or tingling in the back or legs.
Visual analog scale for pain | Change from baseline at 3 days
  Measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured.
  providing a range of scores from 0-10, the following cut points on the pain VAS have been recommended: no pain (0), mild pain(1-3), moderate pain (4-6), and severe pain (>6).
Counter movement jump | Change from baseline at 3 days
  The countermovement jump (CMJ) is a simple, practical, valid, and very reliable measure of lower-body power.
  As a consequence, it is no surprise that this has become a cornerstone test for many strength and conditioning coaches and sports scientists.
  The CMJ has been shown to be the most reliable measure of lower-body power compared to other jump tests.
  Use My jump 2 APP to measure jump height (unit=cent). <30 cm=the subject was fatigue, >30 cm=the subject was normal.
Y balance test | Change from baseline at 3 days
  The YBT requires the athlete to balance on one leg whilst simultaneously reaching as far as possible with the other leg in three separate directions: anterior, posterolateral, and posteromedial.
  Therefore, this test measures the athlete's strength, stability and balance in various directions.
  The YBT composite score is calculated by summing the 3 reach directions and normalizing the results to the lower limb length, whereas asymmetry is the difference between right and left limb reach (1) - this is explained in greater detail in the scoring system section.
Muscle stiffness | Change from baseline at 3 days
  Use Myoton PRO instrument to test the muscle stiffness. The method of measurement consists of recording damped natural oscillation of soft biological tissue in the form of an acceleration signal and the subsequent simultaneous computation of the parameters of State of Tension, Biomechanical and Viscoelastic properties.
  Damped natural oscillation is induced by an exterior, low force quick-release mechanical impulse under constant pre-load.
  The test muscle : Quadriceps, Hamstring, Gastrocnemius, Tibialis anterior muscle.

CONTACTS AND LOCATIONS:
Overall Officials: Wu Chia-Wen, Postgraduate, Principal Investigator — Kaohsiung Medical University Chung-Ho Memorial Hospital
Locations (1):
- Kaohsiung Medical University, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No